CLINICAL TRIAL: NCT00251186
Title: Phase II Study of First-Line Capecitabine and Cetuximab for Treatment of Metastatic Colorectal Cancer in Elderly Patients and/or Those With Multiple Comorbidities Unable to Receive Chemotherapy Doublets
Brief Title: First-Line Capecitabine and Cetuximab for Metastatic Colorectal Ca in Elderly Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding unavailable
Sponsor: University of Medicine and Dentistry of New Jersey (Other)
Collaborators: Rutgers Cancer Institute of New Jersey (Other); Bristol-Myers Squibb (Industry)
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5536; CINJ 070502
Record Dates: First submitted 2005-11-07; First posted 2005-11-09 (Estimated); Last update posted 2010-01-26 (Estimated); Status verified 2010-01

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Capecitabine; Cetuximab

INTERVENTIONS:
Drug: Capecitabine and Cetuximab

SUMMARY:
This is a Phase II clinical trial measuring the effectiveness of the combination of Capecitabine and cetuximab for first line treatment of colorectal cancer in elderly patients and/or those with multiple comorbidities unable to receive standard chemotherapy. This study will be open approximately 2-3 years. Approximately 36 patients will be enrolled on this study. The study will begin enrolling at The Cancer Institute of New Jersey, with 17 patients in the first group. If more than 4 responses are noted, the accrual will continue to 36 patients throughout CINJOG.

ELIGIBILITY:
Inclusion Criteria

* Histologically or cytologically proven diagnosis of locally extensive or metastatic colorectal cancer, not amenable to curative therapy.
* No prior therapy for metastatic disease. Only 5-fluorouracil and leucovorin chemotherapy in the adjuvant setting will be allowed and the last treatment was given more then 6 months prior to metastatic disease development.
* Patients with an ECOG performance score of 2 AND/OR Charlson comorbidity index of ³ 4.
* Patients must be documented by the physician to be medically unable to tolerate oxaliplatin and/or irinotecan based chemotherapy.
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as ³ 20 mm with conventional techniques or as ³10 mm with spiral CT scan.
* Life expectancy of greater than 3 months.
* Laboratory values showing adequate organ function prior to going on-study:

  * Absolute neutrophil count (ANC) ≥ 2.5 x 109/L
  * Platelets (PLT) 100 x 109/L
  * Hemoglobin 9g/dl (with or without transfusion)
  * Metabolic:Calculated creatinine clearance > 50 ml/min
  * Total Bilirubin £ 1.5 x Upper limit of normal (ULN)
  * AST £ 3 x ULN
* Patient should be able to ingest oral medication.
* Ability to understand and sign an approved informed consent.

Exclusion Criteria

* Patients with uncontrolled systemic disease other than the patient's colorectal cancer (e.g., unstable or uncompensated respiratory, cardiac, hepatic, or renal disease) for which the patient was admitted to the hospital within the prior month. Patients with stable respiratory, cardiac, hepatic or renal disease may participate subject to the guidelines in the eligibility criteria above.
* Presence of dementia or delirium.
* Unable to eat, dress, bathe or use the toilet independently. The patient must be able to ambulate independently unless limited by arthritis or musculoskeletal condition.
* Patients with active gastritis within the last 3 months prior to study entry.
* No synchronous or prior malignancy other than non-melanomatous skin cancer or insitu carcinoma of the cervix, unless disease free > 3 years.
* Known dihydropyrimidine dehydrogenase (DPD) deficiency.
* Pregnant women are ineligible as treatment involves unforeseeable risks to the participant and to the embryo or fetus. Women must either be not of child bearing potential or have a negative pregnancy test within 7 days of treatment. Patients are considered not of child bearing potential if they are surgically sterile (they have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or they are postmenopausal. Men and women must be willing to use adequate birth control measures to prevent contraception.
* Inability to or unwillingness to comply with protocol defined treatment and assessments.
* Prior therapy that specifically and directly targets the EGFR pathway.
* Prior severe infusion reaction to a monoclonal antibody.
* Any concurrent chemotherapy not indicated in the study protocol or any other investigational agent(s).
* Patients ingesting herbal supplements, botanicals or vitamins in excess of recommended daily dose must be willing to stop their use, 1 week prior to study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18
Dates: Start 2006-04; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Primary Objective
To measure the response (CR/PR) for a novel chemotherapy/biologic combination-capecitabine/cetuximab for patients with metastatic colorectal cancer who are too fragile for more intensive chemotherapy doublet regimens.

SECONDARY OUTCOMES:
Secondary Objectives
To measure progression-free survival and document overall survival in this patient population.
To assess the toxicity of capecitabine/cetuximab
To describe the baseline quality of life and functional characteristics of elderly patients or those with multiple comorbidities enrolled in this study and assess the impact of disease and its treatment on such functional characteristics.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Poplin, MD, Principal Investigator — Rutgers, The State University of New Jersey
Locations (1):
- The Cancer Institute of New Jersey, New Brunswick, New Jersey, United States